CLINICAL TRIAL: NCT03214016
Title: Effects of Pilates Method and Aerobic Training in Hypertensive Subjects: a Randomized Trial
Brief Title: Effects of Pilates Method and Aerobic Training in Hypertensive Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Santa Maria (Other)
Responsible Party: Principal Investigator, Prof. Dr. Antônio Marcos Vargas da Silva, Physiotherapy professor, Universidade Federal de Santa Maria
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EPMAT
Record Dates: First submitted 2017-07-03; First posted 2017-07-11 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Hypertension
Keywords: Pilates Training; Aerobic Exercises; Hypertension; Clinical trial
MeSH Terms: conditions — Hypertension | interventions — Exercise; Exercise Movement Techniques

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilates method group (Experimental): The participants will do Mat Pilates.
  Interventions: Other: Pilates
- Aerobic training group (Active Comparator): The participants will do aerobic exercise on treadmill.
  Interventions: Other: Aerobic Exercise

INTERVENTIONS:
Other: Aerobic Exercise — 1 hour of aerobic training on a treadmill, 3 times a week, during 8 weeks.
  Other Names: aerobic training
  Arms: Aerobic training group
Other: Pilates — 1 hour of Mat Pilates, 2 times a week, during 8 weeks.
  Other Names: Pilates method; Mat Pilates
  Arms: Pilates method group

SUMMARY:
This study evaluates the effects of Pilates method and aerobic training in hypertensive subjects. Half of participants will be trained with Pilates, while the other half will be trained with aerobic exercise during 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* subjects with high blood pressure controled by medication;
* sedentary.

Exclusion Criteria:

* IMC≥30 kg/m²
* using beta blockers
* smokers or that interrupted the routine less than 6 months
* musculoskeletal diseases in evolution or with current symptomatic
* rheumatological diseases
* other cardiovascular disease
* renal disease due to hypertension
* endocrine, neurological, oncological, immunological, hematological and psychiatric diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-08-20 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline casual systolic blood pressure at 8 weeks | baseline and 8 weeks
  It will be evaluated with oscillometric method of measuring blood pressure with an automated cuff.
Change from baseline 24-hour systolic blood pressure at 8 weeks | baseline and 8 weeks
  It will be evaluated by 24-hour ambulatory BP monitoring (ABPM)

SECONDARY OUTCOMES:
Casual diastolic blood pressure | baseline and 8 weeks
  It will be evaluated with oscillometric method of measuring blood pressure with an automated cuff.
Heart rate variability | baseline and 8 weeks
  It will be evaluated using a previously validated heart rate monitor Polar 810i, and the results will be analyzed in time- and frequency-domains.
Diastolic and mean blood pressure | baseline and 8 weeks
  It will be evaluated by 24-hour ambulatory BP monitoring (ABPM)
Functional capacity | baseline and 8 weeks
  Evaluate by Six-Minute Walk Test (6MWT)
Respiratory muscle strength | baseline and 8 weeks
  The maximal inspiratory and expiratory pressures will be evaluated with manovacuometer
Muscle strength | baseline and 8 weeks
  The muscles (quadriceps, gastrocnemius, abdominal and spine extensors) will be evaluated with dynamometer.
Flexibility | baseline and 8 weeks
  It will be evaluated by bank of Wells test.
Body Mass Index | baseline and 8 weeks
  It will be calculated as weight (kg) divided by height squared.
Oxidative damage | baseline and 8 weeks
  It will be evaluated by advanced oxidation protein products (AOPP)
Antioxidant capacity | baseline and 8 weeks
  It will be evaluated by total antioxidant capacity (TAC).
Lipid profile | baseline and 8 weeks
  By blood analysis (LDL, HDL, total cholesterol, glucose and triglycerides).
Endothelial function | baseline and 8 weeks
  By blood analysis (Nitrite measurement/NOx).
Inflammation | baseline and 8 weeks
  It will be evaluated by C-reactive protein in blood analysis
Creatinine | baseline and 8 weeks
  By blood analysis
Lactate | baselina and 8 weeks
  By blood analysis
Creatine kinase | baseline and 8 weeks
  By blood analysis
Questionnaire of Quality of life | baseline and 8 weeks
  It will be evaluated by Mini-questionnaire of Quality of Life in Hypertension (MINICHAL)

CONTACTS AND LOCATIONS:
Locations (1):
- University Federal of Santa Maria, Santa Maria, Rio Grande do Sul, Brazil